CLINICAL TRIAL: NCT00346775
Title: A Randomized, Single-Blind, Cross-Over, Multicenter Study to Validate the Preference Module of the Experience With Allergic Rhinitis Nasal Sprays Questionnaire (EARNS-Q) Administered to Adult Subjects With Seasonal Allergic Rhinitis During a Three-week Cross-over Study
Brief Title: Validation Of Preference Module Of Experience With Allergic Rhinitis Nasal Sprays Questionnaire (EARNS-Q)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FFR105693
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: questionnaire; nasal spray; Seasonal allergic rhinitis; nasal spray questionnaire; allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — Beclomethasone; flunisolide

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Drug: Beclomethasone dipropionate — Beclomethasone dipropionate
Drug: Flunisolide — Flunisolide
  Other Names: Beclomethasone dipropionate

SUMMARY:
The Protocol section needs to be updated using the following text "The main goal of the study was to validate the Preference Module of the EARNS-Q and to test the reliability using Treatment Satisfaction Questionnaire for Medicines (TSQM), a validated questionnaire for determining satisfaction among different treatment. The EARNS-Q is divided into 2 modules, an Experience Module and a Preference Module. The Experience Module includes 28 items, fourteen attribute rating items followed by fourteen importance weighing questions. The Preference Module includes the same items along with preference questions related to each item as well as a global preference question.

ELIGIBILITY:
Inclusion criteria:

* Seasonal allergic rhinitis.
* Nasal allergy symptoms during the spring allergy season.

Exclusion Criteria:

* Prior use of beclomethasone dipropionate or flunisolide.
* Significant concomitant medical conditions.
* Use of corticosteroids.
* Use of allergy and other identified medications during the study.
* Current tobacco use or tobacco use within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2006-06-29 (Actual); Study Completion 2006-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Napa, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: FFR105693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR105693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR105693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR105693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR105693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR105693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR105693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned on 90 participants, male or female aged 18 years or older, diagnosed with seasonal allergic rhinitis (SAR) across 8 investigational sites in the United States (US) from 01 May 2006 to 29 June 2006.
Pre-assignment Details: A total of 97 participants were randomized for the study in a crossover manner in a ratio of 1:1 to one of two blinded treatment groups of 116 microgram (µg) Nasarel or 168 µg Beconase AQ® metered dose nasal spray to be administered twice daily for 1 week. The study consisted of 2 treatment periods of 1 week each and 1 washout period of 7 days.
Groups:
- Beconase Then Nasarel: Participants were administered 168 µg Beconase AQ metered dose nasal spray twice daily for 1 week. After a washout period of 7 days, participants were administered 116 µg Nasarel, metered dose nasal spray twice daily for 1 week.
- Nasarel Then Beconase: Participants were administered 116 µg Nasarel metered dose nasal spray twice daily for 1 week. After a washout period of 7 days, participants were administered 168 µg Beconase AQ, metered dose nasal spray twice daily for 1 week.
Period: Period 1: Intervention Period 1
Arm/Group | Beconase Then Nasarel | Nasarel Then Beconase
Started | 49 | 48
Completed | 44 | 45
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 3 | 2
Not completed — Participant had nasal congestion score<2 | 1 | 0
Period: Period 2: Washout Period (7 Days)
Arm/Group | Beconase Then Nasarel | Nasarel Then Beconase
Started | 44 | 45
Completed | 44 | 45
Not Completed | 0 | 0
Period: Period 3: Intervention Period 2
Arm/Group | Beconase Then Nasarel | Nasarel Then Beconase
Started | 44 | 45
Completed | 44 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Beconase + Nasarel: Participants were administered 168 µg Beconase AQ or 116 µg Nasarel metered dose nasal spray twice daily for 1 week in a sequence of Beconase /Nasarel or Nasarel/Beconase according to a plan of randomization. The two treatment periods were separated by a washout period of 7 days.
Arm/Group | Beconase + Nasarel
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.1 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 74
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Correlations of Experience With Allergic Rhinitis Nasal Sprays Questionnaire (EARNS-Q) Preference Module With Treatment Satisfaction Questionnaire for Medicines (TSQM) Change Scores and Change in Mean Daily Reflective Total Nasal Symptom (rTNSS) Scores
Description: EARNS-Q Preference Module consists of efficacy, sensory perception (SP), device characteristic (DC), spray delivery (SD), overall product preference (OPP) and total domain. TSQM consists of global satisfaction (GS), convenience, effectiveness and side-effects (SE) domains. Positive (+ve) correlation of EARNS-Q preference scores with change on TSQM domains indicate that preference for a product is associated with better TSQM scores. Negative (-ve) correlation with mean daily rTNSS indicate that preference for a product is associated with lower mean daily rTNSS. Change in TSQM domain scores and mean daily rTNSS was calculated as scores in Treatment Period (TP) 2 minus scores in TP1; change in TSQM is +ve, product in TP2 is preferred, vice-versa; change in rTNSS is -ve, product administered in TP2 is preferred, vice-versa.
Time Frame: Day 1 to Day 23
Population: Intent- to- Treat (ITT) Population was defined as all the participants who were randomized to the study drug. Pearson correlations was used in correlational analyses.
Measure: Number; unit: correlation coefficient
Groups:
- Beconase + Nasarel: Participants were administered 168 µg Beconase AQ or 116 µg Nasarel metered dose nasal spray twice daily for 1 week in a sequence of Beconase /Nasarel or Nasarel/Beconase according to a plan of randomization. The two treatment periods were separated by a washout period of 7 days. After completing TP2, at Visit 5 (Day 22), participants were administered the Preference Module of the EARNS-Q. The TSQM questionnaire was administered to participants at Visits 3 (Day 8) after completion of TP1 and on Visit 5 (Day 22), after completion of TP2. The validity of the Preference Module of the EARNS-Q was assessed by the correlation analysis with change scores (score of TP2 minus scores of TP1) of TSQM questionnaire and rTNSS. Because study medication was changed only once, there was only one assessment of the Preference Module of the EARNS-Q.
Arm/Group | Beconase + Nasarel
Number analyzed (Participants) | 97
correlation coefficient
  EARNS-Q Total-TSQM GS | 0.45
  EARNS-Q Total-TSQM Convenience | 0.45
  EARNS-Q Total-TSQM Effectiveness | 0.44
  EARNS-Q Total-TSQM SE | 0.36
  EARNS-Q Total-Mean rTNSS | -0.39
  EARNS-Q Efficacy-TSQM GS | 0.56
  EARNS-Q Efficacy -TSQM Convenience | 0.30
  EARNS-Q Efficacy-TSQM Effectiveness | 0.59
  EARNS-Q Efficacy -TSQM SE | 0.26
  EARNS-Q Efficacy-Mean rTNSS | -0.53
  EARNS-Q SP-TSQM GS | 0.33
  EARNS-Q SP-TSQM Convenience | 0.38
  EARNS-Q SP-TSQM Effectiveness | 0.33
  EARNS-Q SP-TSQM SE | 0.37
  EARNS-Q SP-Mean rTNSS | -0.27
  EARNS-Q DC-TSQM GS | 0.29
  EARNS-Q DC-TSQM Convenience | 0.49
  EARNS-Q DC-TSQM Effectiveness | 0.24
  EARNS-Q DC-TSQM SE | 0.26
  EARNS-Q DC-Mean rTNSS | -0.21
  EARNS-Q SD-TSQM GS | 0.34
  EARNS-Q SD-TSQM Convenience | 0.37
  EARNS-Q SD-TSQM Effectiveness | 0.30
  EARNS-Q SD-TSQM SE | 0.25
  EARNS-Q SD-Mean rTNSS | -0.27
  EARNS-Q OPP-TSQM GS | 0.54
  EARNS-Q OPP-TSQM Convenience | 0.35
  EARNS-Q OPP-TSQM Effectiveness | 0.52
  EARNS-Q OPP-TSQM SE | 0.30
  EARNS-Q OPP-Mean rTNSS | -0.50

2. Primary Outcome: Correlation of EARNS-Q Preference Module With EARNS-Q Experience Module Change Scores
Description: The 28 items of the EARNS-Q experience module assess 14 attributes with regard to their product rating and their importance of efficacy, SP, DC and SD. The EARNS-Q preference module consists of additional 15 items that evaluate preference by comparing two products based on the same 14 experience attributes as well as on OPP. Change in EARNS-Q Experience Module domain scores was calculated as scores in TP2 minus scores in TP1. If the change in EARNS-Q Experience Module domain scores is +ve, product in TP2 is preferred and vice-versa. A higher product rating for one of the sprays lead to a preference for that spray. The EARNS-Q preference module was assessed only once, at the end of TP2. Positive correlations indicate agreement (i.e. preference for a product is positively associated with better experience with same product).
Time Frame: Day 1 to Day 23
Population: ITT Population. Pearson correlations was used in correlational analyses.
Measure: Number; unit: correlation coefficient
Groups:
- Beconase + Nasarel: Participants were administered 168 µg Beconase AQ or 116 µg Nasarel metered dose nasal spray twice daily for 1 week in a sequence of Beconase /Nasarel or Nasarel/Beconase according to a plan of randomization. The two treatment periods were separated by a washout period of 7 days. After completing TP2, at Visit 5 (Day 22), participants were administered the Preference Module of the EARNS-Q. The Experience Module of EARNS-Q questionnaire was administered on Visit 2 (Day 1) of each TP. The validity of the Preference Module of the EARNS-Q was assessed by the correlation analysis with change scores (score of TP2 minus scores of TP1) of the Experience Module of EARNS-Q questionnaire. Because study medication was changed only once, there was only one assessment of the Preference Module of the EARNS-Q.
Arm/Group | Beconase + Nasarel
Number analyzed (Participants) | 97
correlation coefficient
  Preference Total-Experience Total | 0.72
  Preference Total-Experience Efficacy | 0.38
  Preference Total-Experience SP | 0.66
  Preference Total-Experience DC | 0.42
  Preference Total- Experience SD | 0.38
  Preference Efficacy- Experience Total | 0.47
  Preference Efficacy- Experience Efficacy | 0.55
  Preference Efficacy- Experience SP | 0.29
  Preference Efficacy- Experience DC | 0.20
  Preference Efficacy- Experience SD | 0.29
  Preference SP- Experience Total | 0.75
  Preference SP - Experience Efficacy | 0.25
  Preference SP - Experience SP | 0.79
  Preference SP - Experience DC | 0.43
  Preference SP - Experience SD | 0.29
  Preference DC- Experience Total | 0.63
  Preference DC - Experience Efficacy | 0.20
  Preference DC - Experience SP | 0.59
  Preference DC - Experience DC | 0.45
  Preference DC- Experience SD | 0.38
  Preference SD- Experience Total | 0.47
  Preference SD - Experience Efficacy | 0.24
  Preference SD - Experience SP | 0.38
  Preference SD - Experience DC | 0.32
  Preference SD- Experience SD | 0.39
  Preference OPP- Experience Total | 0.59
  Preference OPP - Experience Efficacy | 0.44
  Preference OPP - Experience SP | 0.47
  Preference OPP - Experience DC | 0.33
  Preference OPP- Experience SD | 0.35

3. Secondary Outcome: Mean rTNSS Over Period
Description: The rTNSS score is the sum of the four individual symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing. Each symptom is scored on a 4 point scale ranging from 0 to 3. Each individual symptom was evaluated using a scale of 0 (none; symptom is not present), 1 (mild; sign/symptom clearly present but minimal awareness; easily tolerated), 2 (moderate; definite awareness of sign/symptom that is bothersome but tolerable), or 3 (severe; sign/symptom is hard to tolerate; causes interference with activities of daily living and/or sleeping). The rTNSS ranges from 0 (none) to 12 (severe). Higher score represents greater severity of symptoms. The reflective assessment of the TNSS scores the four nasal symptoms over the previous 12 hours and are assessed in the morning and evening. The participants themselves scored nasal symptoms in a diary card. The analysis was done based on the rTNSS averaged over the two weeks of the treatment period.
Time Frame: Day 1 to 8 of each treatment period
Population: Efficacy population was defined as all participants who completed both treatment periods, who had efficacy and questionnaire data recorded in both treatment periods, and who had recorded sufficient efficacy data to calculate daily rTNSS.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Groups:
- Beconase: In each period of the study, participants were administered 168 µg Beconase AQ metered dose nasal spray twice daily for 1 week according to a plan of randomization. The two treatment periods were separated by a washout period of 7 days.
- Nasarel: In each period of the study, participants were administered 116 µg Nasarel metered dose nasal spray twice daily for 1 week according to a plan of randomization. The two treatment periods were separated by a washout period of 7 days.
Arm/Group | Beconase | Nasarel
Number analyzed (Participants) | 89 | 89
Score on scale | 5.3 (0.28) | 5.1 (0.28)
Statistical Analysis 1: Comparison: Beconase vs Nasarel; Test type: Superiority or Other; p = 0.517, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.6 to 0.3]

4. Secondary Outcome: Number or Participants With Preference of Nasal Sprays (Nasarel or Beconase AQ) at the End of the Last Cross-over Period Using the Preference Module of the EARNS-Q
Description: The participants with preference of nasal sprays (Nasarel or Beconase AQ) at the end of the last cross-over period was planned to be analyzed using the preference module of the EARNS-Q. The data for this outcome measure was not collected and the result summary was not generated.
Time Frame: Up to Day 23
Population: Efficacy Population. No participants were analyzed for this outcome measure.
Groups:
- Beconase: In each period of the study, participants were administered 168 μg Beconase AQ metered dose nasal spray twice daily for 1 week according to a plan of randomization. The two treatment periods were separated by a washout period of 7 days.
- Nasarel: In each period of the study, participants were administered 116 μg Nasarel metered dose nasal spray twice daily for 1 week according to a plan of randomization. The two treatment periods were separated by a washout period of 7 days.
Arm/Group | Beconase | Nasarel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Post randomization (Day 1) up to 23 days
Description: ITT Population was used for analysis.
Arm/Group | Beconase | Nasarel
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/97
Other Adverse Events (participants affected / at risk) | 16/97 | 17/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Beconase (N=97) | Nasarel (N=97)
Headache (Nervous system disorders) | 7 | 9
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eye infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Hangover (General disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.